CLINICAL TRIAL: NCT01600508
Title: . A Randomized Controlled Trial Comparing Videoconference and Outpatient Stoma Care
Brief Title: Videoconference in Stoma Out-patient Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/1432a (REK)
Record Dates: First submitted 2012-04-03; First posted 2012-05-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Surgical Operation With Formation of External Stoma
Keywords: stoma care; videoconference; costs; quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional stoma care (Active Comparator): Being discharged from a hospital with a stoma is a challenge to the patient's quality of life in many aspects. Optimal stoma function and care is essential to keep quality of life best possible. Videoconference can be a useful tool to help patients cope with stoma problems without travelling long distances to a surgical outpatient clinic.
  Interventions: Other: Videoconference stoma care
- Videoconference Stoma Consultations (Experimental): Videoconference Stoma Consultations
  Interventions: Other: Videoconference stoma care

INTERVENTIONS:
Other: Videoconference stoma care — Stoma patients are randomized to videoconference stoma care or surgical outpatients clinic stoma care

SUMMARY:
Background:

Videoconference (VC) is a common clinical tool and has huge potential to alter medical practice and to offer patients the best expertise in treatment and follow-up in spite of long distances, especially in rural areas. Studies upon selected patient groups have shown that VC is safe and cost-effective. However, RCT of VC patients with stoma problems have never been performed.

Patients with stoma problems are resource demanding patients. The University Hospital North Norway (UNN) has several hundred consultations for this patient group each year, serving the population in North Norway.

Methods: In this randomised controlled trial (RCT), patients are either randomised to a VC consultation or a regular consultation at the outpatient clinic. All patients with a stoma that needs special attention are eligible for inclusion. Patients randomised to the VC group, are set-up to a meeting at the nearest VC studio located to their home community. There will be educated VC- stoma nurses that will participate in the clinical examination at the hospital outpatient clinic and at the rural VC studio.

Endpoints: Primary endpoints are patient satisfaction and quality of life. Secondary endpoints are number of consultations and cost effectiveness.

Sample size calculations showed that 170 patients had to be included in the trial.

The investigators hypothesize that postoperative follow-up of stoma patients by VC will not have any impact on patients' quality of life compared to Hospital outpatient follow-up. Furthermore, the investigators hypothesize that the incremental cost-effectiveness ratio will improve.

DETAILED DESCRIPTION:
There has been substantial development in the uses of VC among medical personnel [1]. Therefore, new applications of VC are emerging, such as surgical telementoring, trauma and emergency medicine, postoperative follow-up of patients, education of medical personnel, and multidisciplinary team meetings [2]. VC has a great and unused potential, this is recently described in an "invited commentary" in World Journal of Surgery [3]. Furthermore, during recent years, the cost of VC equipment has become less expensive, and advanced technical skills are not required to use the system.

Patients with stoma problems are a large and resource demanding group. Each year there are performed several hundred consultations at the surgical outpatient clinic at University Hospital of North-Norway for this patient group. These patients are surgically treated at the gastrointestinal, urological and gynaecological department.

The visual component is critical to give patients with stoma problems the best care, VC will therefore be well suited for this patient group [4, 5]. Furthermore, the infrastructure for VC in northern Norway is well developed for VC. In the county of Finnmark, Troms and Nordland there are a VC network, all linked together through the Norwegian Health Network.

The purpose of this study is to obtain insight into quality of life (QoL) among patients followed up in a hospital outpatient setting or by VC, and into the incremental cost-effectiveness ratio from the point of view of health care and of society.

Methods and design Study design This study is a randomized controlled trial where patients either will be randomized to follow up at the surgical outpatient clinic (control group) or by VC (intervention group

Participants Patients (inclusion and exclusion criteria's)

Medical doctors

Stoma nurses

Intervention Patients are randomized to follow-up either by VC (intervention) or at the surgical outpatient clinic. All patients will receive their first postoperative check-up at the hospital. A clinical examination will then be performed and information about the RCT given. If the patient gives informed consent, randomization is performed. Patients randomized to VC follow-up are referred to their GP and the local VC stoma nurse.

Control arm Patients in the control group consist of patients randomized to regular follow-up at the hospital's surgical outpatient clinic. This follow-up is performed by consultants in digestive surgery, or a specially educated stoma nurse. QOL questionnaires The EQ-5D questionnaires for the two-year follow-up period (at 1, 3, 6, 9, 12, 15, 18, 21, 24 month follow-up) are given to the patient at baseline examination. Economic evaluation questionnaire: A questionnaire has been developed to enable calculation of costs related to patient examinations. This questionnaire is incorporated in the QOL questionnaire, and patients are requested to fill out the questionnaire at 1, 3 6, 9, 12, 15, 18, 21 and 24 months after inclusion. The cost elements will include patient- and family-related costs due to outpatient visits, VC visits, laboratory tests, radiographs/ultrasound, examinations due to stoma complications, treatment of stoma complications, traveling, production losses, co-payments and other patient expenses. Control arm Patients in the control group consist of patients randomized to regular follow-up at the hospital's surgical outpatient clinic. Consultants in digestive surgery or stoma nurses perform this follow-up.

Objectives Primary objective We aim to compare quality of life and costs of follow-up among patients followed up by VC or at the surgical outpatient clinic. We hypothesize that patients followed up by VC will experience similar or higher scores on quality of life measures and lower costs during follow-up.

Secondary objective We want to establish a nurse led VC stoma school, prior to the clinical trial. Nurses, specially educated to treat patient with stoma problems, will write the curriculum. Five to ten nurses from logistic important VC communities all over North Norway will be invited to a 10 to 20 hour course in stoma treatment and technical aspects around VC. This will be done prior to the start of the clinical study.

Outcome measures Primary outcome (measured at 1, 3, 6,9,12,15,18,21 and 24 months) Quality of life EQ-5D is a standardized generic instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status.

EQ-5D measures five dimensions of health-related quality of life (HRQOL): mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ Visual Analogue Scale: The EQ VAS records the respondent's self-rated health status on a vertically graduated (0-100) visual analogue scale [6]. Economic analysis A cost-effectiveness analysis will be performed alongside the randomized controlled trial. A Markov model will be employed. If the trial reveals no difference in health outcomes or quality of life of the patients, a cost-minimization analysis will be carried out. If we reveal a difference in quality of life between the two groups, we will implement a cost-utility analysis. The economic evaluation will have a health care and societal perspective. Resources used in both treatment arms will be registered prospectively based on reports by the patients and on the hospital patient records. Costs related to consultations at the primary and secondary care level, both at baseline and up to 24 months after randomization, including direct medical costs, indirect costs (production losses), travel costs and patient-/family-related costs will be registered. Quality of life measurements will be collected both at baseline and at several time points during the intervention. A 3% discount rate will be used to discount future costs and benefits.

The cost elements will include costs related to outpatient visits, GP visits, laboratory tests, radiographs and ultrasound, examinations due to suspected stoma complications, treatment of stoma complications, traveling/transportation, and production losses, co-payments and other patient/family expenses. The net costs and outcomes of the two treatment options will be compared and presented as incremental cost-effectiveness ratios.

Sample size Sample size calculations are according to Campbell's [7] and EQ-5D guidelines [8]. Alpha and beta were set at 0.05 and 0.2 respectively and tests were two-sided. We hypothesize that patients followed up by VC will have a minor to moderate increase in the QoL scores. Allowing for a dropout rate of 20%, detecting this difference with confidence we required a total sample size of 170 patients.

Randomization Randomization will be done at the 1-month check-up (baseline) after the patients have given informed consent. The randomization service is web-based and managed by the Norwegian University of Science and Technology.

Patients allocated to VC follow-up may be referred back to surgical clinics at any point in the study. Data gathering Data are being collected for patients in the intervention and the control group in identical ways. QoL and "cost questionnaires" are sent after each follow-up appointment by the patients to the trial center up to 24 months postoperatively. These questionnaires are optically readable, data being consecutively collected in a trial database. SCEs are registered via hospital chart review at 24 months postoperatively. The Norwegian Data Inspectorate has approved the study. All data will be handled with strict confidentiality, and study reports or presentations will maintain the anonymity of patients, surgeons, GPs and hospitals. Data collection will be complete by the end of 2013.

Analysis We will use the intention-to-treat principle when analyzing data. Treatment arms will be compared with respect to potential covariates using continuous and categorical univariable analyses. These will include variables relating to patients (age, sex, comorbidities, cost), treatment (surgical resection, surgical complications), hospital surgical outpatient clinic (cost, patient satisfaction, QoL), VC consultation (cost, patient satisfaction, QoL). The cost elements will include costs related to outpatient visits, VC visits, laboratory tests, radiographs/ultrasound, and examinations due to suspected complications, treatment of complications, traveling/transportation, production losses, co-payments and other patient expenses. The net costs and outcomes of the two treatment/follow-up options will be compared and presented as cost-effectiveness ratios. If the trial reveals no difference in health outcomes or quality of life for the patients, a cost-minimization analysis will be carried out. If we find a difference in quality of life or overall survival rates between the two groups, we will use a cost utility approach. The economic evaluation will have a societal and health care perspective. The method of analysis, including adjusting for covariates will comply with the CONSORT statement [9]. The results will be expressed as odds ratios for binary outcomes, hazard ratios for time- to-event outcomes or mean differences for continuous outcomes with corresponding standard errors, 95% confidence intervals, and associated p-values. P-values will be reported to three decimal places with p-values less than 0.001 reported as p < 0.001. For all tests we will use alpha = 0.05 level of significance.

Ethics The Regional Committee for Medical Research Ethics, North Norway approved this protocol. Patients must provide written consent before entering the trial.

Discussion VC is used as an instrument for follow-up of patients in the postoperative period and for outpatient consultation. From our hospital, we have extensive experience in the use of VC in the follow-up of haemodialysis patients [10] and in dermatology [11, 12]. In addition, a new project has started in the orthopaedic department, where a VC line has been established between the University Hospital and the district medical centre Nordreisa, 155 miles away. In this project, both outpatient patients and postoperative patients are examined by a district orthopaedic nurse under the supervision of an orthopaedic consultant located at the University Hospital. This project has now been organized as a randomised controlled trial, where the primary endpoints are cost-effectiveness and patient satisfaction.

Several articles have reported the use of VC in the follow-up of surgical patients. Wallace et al. aimed to compare joint VC between general practitioners, specialists (surgeons), and patients with standard outpatient referral. This randomised controlled trial showed that allocation of patients to virtual outreach consultations was variably associated with increased offers of follow-up appointments according to site and specialty, but led to significant increases in patients' satisfaction and substantial reductions in tests and investigations. Efficient operation of such services will require appropriate selection of patients, significant service reorganization, and provision of logistical support [13].

A study from Finland investigated the use of VC in the examination of orthopaedic outpatients. VC was found to be feasible and the equipment functioned well technically. The conclusion was that VC between primary and secondary care could be used in the examination of orthopaedic patients whenever no demanding imaging technology was needed [14] Whether VC is cost-effective in the follow-up of surgical patients is debated. The clinical effectiveness and costs of VC in orthopaedics between primary and secondary care were examined in an eight-month prospective comparative study. The general surgery outpatient clinics of two Finnish district hospitals were compared. The direct costs of an outpatient visit were 45% greater per patient than for a VC. A cost-minimization analysis of the alternative interventions showed a net benefit of EU 2,500 in favour of VC [15].

Another Finnish study had similar results. Wider utilization of the VC equipment for other purposes, or the use of less expensive VC equipment, would make services cost saving even at relatively short distances [16].

VC can be used in almost any medical specialty, although the specialties best suited are those with a high visual component. Wound healing and wound management are thus prime candidates for VC follow-up. Development of a suitable telemedical system in this field could have a significant effect on wound care in the community, tertiary referral patterns, and hospital admission rates [5, 17].

ELIGIBILITY:
Inclusion Criteria:

* Stoma patients

Exclusion Criteria:

* Not able to travel,
* Accepted written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life | up to two years
  We aim to compare quality of life measured with EQ-5D questionnaires among patients followed up by VC vs those followed up at the surgical outpatient clinic at 1, 3, 6, 9, 12, 15, 18, 21, 24 months of follow-up. We hypothesize that patients followed up by VC will experience similar or higher scores on quality of life measures during followup.

SECONDARY OUTCOMES:
Cost effectiveness | up to two years
  Economic evaluation questionnaire, incorporated in the QOL questionnaire, is given to the patients and requested to fill out at baseline and at 1, 3 6, 9, 12, 15, 18, 21 and 24 months after inclusion. It has been developed to enable calculation of costs related to patient examinations such as patient- and family-related costs due to outpatient visits, VC visits, laboratory tests, radiographs/ultrasound, examinations due stoma complications, treatment of complications, traveling, production losses, co-payments and other patient expenses.

CONTACTS AND LOCATIONS:
Overall Officials: Rolv-Ole Lindsetmo, MD, PhD, MPH, Principal Investigator — Institute of Clinical Medicine, Tromsø University, Norway, Univertsity Hospital of North Norway

REFERENCES:
- [Background] Jarvis-Selinger S, Chan E, Payne R, Plohman K, Ho K. Clinical telehealth across the disciplines: lessons learned. Telemed J E Health. 2008 Sep;14(7):720-5. doi: 10.1089/tmj.2007.0108. PMID 18817503
- [Background] Augestad KM, Lindsetmo RO. Overcoming distance: video-conferencing as a clinical and educational tool among surgeons. World J Surg. 2009 Jul;33(7):1356-65. doi: 10.1007/s00268-009-0036-0. PMID 19384459
- [Background] Doarn CR. The power of video conferencing in surgical practice and education. World J Surg. 2009 Jul;33(7):1366-7. doi: 10.1007/s00268-009-0042-2. No abstract available. PMID 19390758
- [Background] Shannon RJ. Telemedicine in wound healing. Int Wound J. 2005 Sep;2(3):239-40. doi: 10.1111/j.1742-4801.2005.0124b.x. No abstract available. PMID 16618327
- [Background] Wilbright WA, Birke JA, Patout CA, Varnado M, Horswell R. The use of telemedicine in the management of diabetes-related foot ulceration: a pilot study. Adv Skin Wound Care. 2004 Jun;17(5 Pt 1):232-8. doi: 10.1097/00129334-200406000-00012. PMID 15192491
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Campbell MJ, Julious SA, Altman DG. Estimating sample sizes for binary, ordered categorical, and continuous outcomes in two group comparisons. BMJ. 1995 Oct 28;311(7013):1145-8. doi: 10.1136/bmj.311.7013.1145. PMID 7580713
- [Background] Roset M, Badia X, Mayo NE. Sample size calculations in studies using the EuroQol 5D. Qual Life Res. 1999 Sep;8(6):539-49. doi: 10.1023/a:1008973731515. PMID 10548869
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066
- [Background] Rumpsfeld M, Arild E, Norum J, Breivik E. Telemedicine in haemodialysis: a university department and two remote satellites linked together as one common workplace. J Telemed Telecare. 2005;11(5):251-5. doi: 10.1258/1357633054471885. PMID 16035968
- [Background] Moseng D. [Teledermatology--experiences from Northern Norway]. Tidsskr Nor Laegeforen. 2000 Jun 20;120(16):1893-5. Norwegian. PMID 10925620
- [Background] Nordal EJ, Moseng D, Kvammen B, Lochen ML. A comparative study of teleconsultations versus face-to-face consultations. J Telemed Telecare. 2001;7(5):257-65. doi: 10.1258/1357633011936507. PMID 11571079
- [Background] Wallace P, Haines A, Harrison R, Barber J, Thompson S, Jacklin P, Roberts J, Lewis L, Wainwright P; Virtual Outreach Project Group. Joint teleconsultations (virtual outreach) versus standard outpatient appointments for patients referred by their general practitioner for a specialist opinion: a randomised trial. Lancet. 2002 Jun 8;359(9322):1961-8. doi: 10.1016/s0140-6736(02)08828-1. PMID 12076550
- [Background] Haukipuro K, Ohinmaa A, Winblad I, Linden T, Vuolio S. The feasibility of telemedicine for orthopaedic outpatient clinics--a randomized controlled trial. J Telemed Telecare. 2000;6(4):193-8. doi: 10.1258/1357633001935347. PMID 11027118
- [Background] Harno K, Arajarvi E, Paavola T, Carlson C, Viikinkoski P. Clinical effectiveness and cost analysis of patient referral by videoconferencing in orthopaedics. J Telemed Telecare. 2001;7(4):219-25. doi: 10.1258/1357633011936435. PMID 11506757
- [Background] Ohinmaa A, Vuolio S, Haukipuro K, Winblad I. A cost-minimization analysis of orthopaedic consultations using videoconferencing in comparison with conventional consulting. J Telemed Telecare. 2002;8(5):283-9. doi: 10.1177/1357633X0200800507. PMID 12396857
- [Background] Jones SM, Banwell PE, Shakespeare PG. Telemedicine in wound healing. Int Wound J. 2004 Dec;1(4):225-30. doi: 10.1111/j.1742-4801.2004.00055.x. PMID 16722871
- [Derived] Augestad KM, Sneve AM, Lindsetmo RO. Telemedicine in postoperative follow-up of STOMa PAtients: a randomized clinical trial (the STOMPA trial). Br J Surg. 2020 Apr;107(5):509-518. doi: 10.1002/bjs.11491. Epub 2020 Feb 26. PMID 32100297